CLINICAL TRIAL: NCT03394638
Title: Assessing the Value of eHealth for Bariatric Surgery
Acronym: BePATIENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Dirk Versteegden, MD, Catharina Ziekenhuis Eindhoven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL56992.100.16
Record Dates: First submitted 2017-12-06; First posted 2018-01-09 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Bariatric Surgery; Obesity; Telemedicine
Keywords: eHealth; Bariatric surgery; Obesity; Telemedicine
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional group (Active Comparator): Treatment includes:
  1. 10 individual and 3 group consultations at the outpatient department by several disciplines in the first postoperative year.
  2. Additional visits if necessary
  3. No further access to the BePATIENT website
  Interventions: Procedure: Conventional group
- Online group (Experimental): Treatment includes:
  Added to conventional group: Continuation of access to the BePATIENT website with:
  1. eLearning programs
  2. Informative videos
  3. Patient network
  4. Video consulting
  Interventions: Other: Access to online eLearning module; Procedure: Conventional group
- Device group (Experimental): Added to Online group:Four wireless devices, which are
  1. Weight Scale
  2. Blood Pressure
  3. Oximeter
  4. Activity Tracker
  Interventions: Other: Access to online eLearning module; Other: Access to measurement devices; Procedure: Conventional group

INTERVENTIONS:
Other: Access to online eLearning module — Patients enrolled in the Online group have access to an online platform called BePatient. Patients are given the ability to access the platform and do eLearnings; watch videos about the operation and recovery; do quizzes, see dietary advices; see news about obesity and our department; read patients' stories. They are also able to chat with other patients.
  Arms: Device group; Online group
Other: Access to measurement devices — Patients in the device group have, in addition to patients in the Online group, access to 4 measuring devices, including: weight scale, oximeter, activity bracelet and blood pressure device. Those devices are connectable to their mobile phones where patients can view their own progress.
  Arms: Device group
Procedure: Conventional group — All patients undergo the standard of care which included: the bariatric procedure and several outpatient visits including consultation with their surgeon, obesity nurses, dieticians and (if indicated) psychologists.

SUMMARY:
Bariatric surgery is the only treatment with long standing effect of morbid obesity. The key elements to success are the patient-selection, an experienced bariatric team and a completed follow-up program. Follow-up programs can consist of, for example, providing social support in support groups, teaching psychological skills, such as coping with the body change or teaching self-regulation of body weight. Furthermore, follow-up is important for dietary and sports counselling. The experience of the team members and coaching skills are essential in indicating the suitable procedure if necessary and guide the patients through the process. Various studies showed a significant positive effect of a completed follow-up program after bariatric surgery on maintaining weight loss. There is a burden for this on site provided care as organizational and financial resources are not unlimited. Especially as the follow-up period is an obligatory 5 years or if possible life long. Even if this aftercare is provided, not all patients complete the complete program. Various reasons are possible for an increasing no-show-rate, the loss of enthusiasm for onsite visits could be one of them. Analogue to other chronic diseases, the addition of telehealth could be useful. Telehealth is the delivery of health-related services and information via telecommunications technologies. It encompasses preventative, promotive and curative aspects. Examples are exchanging health services or education via videoconference, transmission of medical data for disease management (remote monitoring) and advice on prevention of diseases and promotion of good health by patient monitoring and follow-up. The participation of eHealth has been investigated and considered useful in the treatment of obesity. In a systematic review self-measured blood pressure monitoring was associated with better control of hypertension at least in the first year. Its value in a bariatric tract has not been investigated. It can be hypothesized that self-control by eHealth could enhance clinical outcome as more weight loss and comorbidity reduction. Long-term realistic goals setting, consistent use of routines and self-monitoring has been proven effective for weight loss maintenance. Patients with higher self-control are more certain regarding their abilities, which cause higher commitment and adherence to the program. This eventually leads to more weight loss. For this purpose an online monitoring program was designed for our Obesity Centre (BePATIENT) to provide preoperative information as well as aids in the post-bariatric phase by self-control wireless devices for registration of biometric outcomes, teleconference opportunities and access to additional information. In a prospective trial the implementation in several degrees is evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Completed the questionnaire online
2. Having ongoing access to internet
3. Ability to use a model of mobile device (smartphone or tablet) with any version of the Android or iOS platform
4. A body mass index above 40 kg/m2 or above 35 kg/m2 with related comorbidity (hypertension, diabetes type 2, hyperlipidaemia, obstructive sleep apnea syndrome or joint arthritis of lower limbs)
5. A primary gastric sleeve or bypass planned
6. Age of 18 years or more
7. Ability to read and write the Dutch language
8. Signed informed consent

Exclusion Criteria:

1. Patients not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-02-21 (Actual); Primary Completion 2019-12-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | 2 years after the operation
  The BMI in kg/m2 at 2 years postoperatively.

SECONDARY OUTCOMES:
Quality of Life | At 1 and 2 years after the operation
  Quality of Life assessment using the RAND36-questionnaire. The RAND36 questionnaire consists of 36 questions about health related quality of life. The RAND36 scores are divided in 9 subscales: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health and health change. Scores for each subscale are transformed to a linear 0 - 100 score. A higher score indicates a better quality of life in that domain.
Evolution of obesity related comorbidities | At 1 and 2 years after the operation
  Status of comorbidities are recorded at 1 and 2 years postoperatively and classified as either: cured (no medication and no complaints), improved (less medication needed and/or less complaints), unchanged (no alterations in medication use and no change in complaints), worsened (more medication needed and/or more complaints) or de novo (development of a comorbidity which was not present at inclusion). The reviewed comorbidities include: hypertension, diabetes mellitus, Arthralgia, obstructive sleep apnea syndrome, dyslipidemia and gastro-esophageal reflux disease.
Program commitment | At 1 and 2 years after the operation
  A 6-item questionnaire to assess program commitment (Neubert & Cady 2001).
Technical errors biometric devices | At 2 years after the operation
  Number of technical issues reported by patients or health care professionals
Length of hospitalization | At 2 years after the operation
  Length of stay in hospital (days)
Return to work (days) | At 1 year after the operation.
  Number of days patients start working again after operation
Patients' satisfaction | At 1 and 2 years after the operation
  Satisfactory assessment patients (Numeric Rate Scale 0-10)
Health care suppliers' satisfaction | At 1 and 2 years after the operation
  Satisfactory assessment health care professional (Numeric Rate Scale 0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Nienhuijs, MD, PhD, Principal Investigator — Department of Surgery, Catharina Hospital Eindhoven
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Livhits M, Mercado C, Yermilov I, Parikh JA, Dutson E, Mehran A, Ko CY, Shekelle PG, Gibbons MM. Is social support associated with greater weight loss after bariatric surgery?: a systematic review. Obes Rev. 2011 Feb;12(2):142-8. doi: 10.1111/j.1467-789X.2010.00720.x. PMID 20158617
- [Background] [2] Lyons K, Meisner B, Sockalingam S, Cassin S.. Body image after bariatric surgery: A qualitative study. Bariatric Surgical Practice and Patient Care. March 2014, 9(1): 41-49.
- [Background] Petasne Nijamkin M, Campa A, Samiri Nijamkin S, Sosa J. Comprehensive behavioral-motivational nutrition education improves depressive symptoms following bariatric surgery: a randomized, controlled trial of obese Hispanic Americans. J Nutr Educ Behav. 2013 Nov-Dec;45(6):620-6. doi: 10.1016/j.jneb.2013.04.264. Epub 2013 Jun 29. PMID 23819903
- [Background] Mundi MS, Lorentz PA, Grothe K, Kellogg TA, Collazo-Clavell ML. Feasibility of Smartphone-Based Education Modules and Ecological Momentary Assessment/Intervention in Pre-bariatric Surgery Patients. Obes Surg. 2015 Oct;25(10):1875-81. doi: 10.1007/s11695-015-1617-7. PMID 25702141
- [Background] Bond DS, Thomas JG. Measurement and Intervention on Physical Activity and Sedentary Behaviours in Bariatric Surgery Patients: Emphasis on Mobile Technology. Eur Eat Disord Rev. 2015 Nov;23(6):470-8. doi: 10.1002/erv.2394. Epub 2015 Sep 2. PMID 26331982
- [Background] Kim HJ, Madan A, Fenton-Lee D. Does patient compliance with follow-up influence weight loss after gastric bypass surgery? A systematic review and meta-analysis. Obes Surg. 2014 Apr;24(4):647-51. doi: 10.1007/s11695-014-1178-1. PMID 24464545
- [Background] Sysko R, Hildebrandt TB, Kaplan S, Brewer SK, Zitsman JL, Devlin MJ. Predictors and correlates of follow-up visit adherence among adolescents receiving laparoscopic adjustable gastric banding. Surg Obes Relat Dis. 2014 Sep-Oct;10(5):914-20. doi: 10.1016/j.soard.2014.03.012. Epub 2014 Mar 28. PMID 25066443
- [Background] Haggerty AF, Huepenbecker S, Sarwer DB, Spitzer J, Raggio G, Chu CS, Ko E, Allison KC. The use of novel technology-based weight loss interventions for obese women with endometrial hyperplasia and cancer. Gynecol Oncol. 2016 Feb;140(2):239-44. doi: 10.1016/j.ygyno.2015.11.033. Epub 2015 Nov 28. PMID 26644265
- [Background] Skoyen JA, Rutledge T, Wiese JA, Woods GN. Evaluation of TeleMOVE: a Telehealth Weight Reduction Intervention for Veterans with Obesity. Ann Behav Med. 2015 Aug;49(4):628-33. doi: 10.1007/s12160-015-9690-7. PMID 25697133
- [Background] Azar KM, Aurora M, Wang EJ, Muzaffar A, Pressman A, Palaniappan LP. Virtual small groups for weight management: an innovative delivery mechanism for evidence-based lifestyle interventions among obese men. Transl Behav Med. 2015 Mar;5(1):37-44. doi: 10.1007/s13142-014-0296-6. PMID 25729451
- [Background] Steinberg DM, Levine EL, Lane I, Askew S, Foley PB, Puleo E, Bennett GG. Adherence to self-monitoring via interactive voice response technology in an eHealth intervention targeting weight gain prevention among Black women: randomized controlled trial. J Med Internet Res. 2014 Apr 29;16(4):e114. doi: 10.2196/jmir.2996. PMID 24780934
- [Background] Luley C, Blaik A, Gotz A, Kicherer F, Kropf S, Isermann B, Stumm G, Westphal S. Weight loss by telemonitoring of nutrition and physical activity in patients with metabolic syndrome for 1 year. J Am Coll Nutr. 2014;33(5):363-74. doi: 10.1080/07315724.2013.875437. Epub 2014 Aug 8. PMID 25105874
- [Background] Ahrendt AD, Kattelmann KK, Rector TS, Maddox DA. The effectiveness of telemedicine for weight management in the MOVE! Program. J Rural Health. 2014 Winter;30(1):113-9. doi: 10.1111/jrh.12049. Epub 2013 Sep 24. PMID 24112223
- [Background] Uhlig K, Patel K, Ip S, Kitsios GD, Balk EM. Self-measured blood pressure monitoring in the management of hypertension: a systematic review and meta-analysis. Ann Intern Med. 2013 Aug 6;159(3):185-94. doi: 10.7326/0003-4819-159-3-201308060-00008. PMID 23922064
- [Background] McKee H, Ntoumanis N, Smith B. Weight maintenance: self-regulatory factors underpinning success and failure. Psychol Health. 2013;28(10):1207-23. doi: 10.1080/08870446.2013.799162. Epub 2013 Jun 14. PMID 23767689
- [Derived] Versteegden DPA, Van Himbeeck MJJ, Luyer MD, van Montfort G, de Zoete JJGM, Smulders JF, Nienhuijs SW. A randomized clinical trial evaluating eHealth in bariatric surgery. Surg Endosc. 2023 Oct;37(10):7625-7633. doi: 10.1007/s00464-023-10211-w. Epub 2023 Jul 20. PMID 37474829